CLINICAL TRIAL: NCT02358603
Title: Investigation of the Chronotropic Incompetence Diagnostic Algorithm in Heart Failure Patients
Brief Title: Chronotropic Incompetence (CI) Diagnostic Algorithm in Heart Failure Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CI in Heart Failure Study
Record Dates: First submitted 2014-05-16; First posted 2015-02-09 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
Keywords: Chronotropic Incompetence; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Case group subjects will complete study required protocol testing while wearing an experimental device, the ActiGraph device placed on his/her wrist and a Holter device with ECG electrodes placed on his/her chest. Results will be compared to a Control Group.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case group (Experimental): At the beginning of the study, each subject of the case group will complete echo examination and related lab test for BNP. During the study, each subject will have a six minutes' walk test and 24 hour ambulatory monitoring while having an ActiGraph device placed on his/her wrist and a Holter device with ECG electrodes placed on his/her chest. The treadmill test is optional to patients per physicians' instruction and/or patients' own judgment. It would be performed at the end of the study if chosen.
  Interventions: Diagnostic Test: Chronotropic Incompetence Diagnostic Algorithm
- Control group (Placebo Comparator): Each subject of the control group will do the same test and examination with the subjects in the case group.
  Interventions: Diagnostic Test: Chronotropic Incompetence Diagnostic Algorithm

INTERVENTIONS:
Diagnostic Test: Chronotropic Incompetence Diagnostic Algorithm
  Other Names: Standard of Care Diagnostic Testing

SUMMARY:
This study is to collect human activity and electrocardiogram (ECG) data from heart failure (HF) patients to aid in the development of a novel chronotropic incompetence (CI) algorithm designed to diagnose CI in patients with HF.

DETAILED DESCRIPTION:
The Investigation of the Chronotropic Incompetence Diagnostic Algorithm in Heart Failure Patients (CI Algorithm Study) is an acute data collection study using market released actigraphy devices (wGT3X-BT) and holter devices (DR 180) to measure study subjects' daily activities and surface ECG data simultaneously. The data will be analyzed to develop an algorithm to diagnose CI in patients with HF.

ELIGIBILITY:
Inclusion criteria for the case group:

* Patient is greater than 18 years of age and less than 70 years of old.
* Patient is willing and able to give informed consent.
* Patient has been diagnosed with stable chronic HF according to European Society of Cardiology 2012 HF guidance.
* New York Heart Association class I- III, including with HF with preserved ejection fraction and HF with reduced ejection fraction patients.
* Patients can perform moderate exercise.
* Left ventricular ejection fraction less than 55% but greater than 35%.

Inclusion criteria for the control group:

* Subject is greater than 18 years of age and less than 70 years of old.
* Subject is willing and able to give informed consent.

Exclusion criteria for the case group:

* Patient is unable or unwilling to sign the patient informed consent.
* Patient has implantable pacemaker, Implantable cardiovert defibrillator (ICD) or cardiac resynchronize therapy (CRT) device.
* Patient has at least one pacemaker, ICD or CRT indications.
* Patients has persistent atrial fibrillation (AF).
* Patient whose hear rate baseline at the rest is greater than 95 beats per minutes (BPM).
* Patient has contraindications for cardio-pulmonary exercise testing, including but not limited to, unstable angina, decompensated heart failure, active pericarditis or myocarditis and ECG ST-segment shift > 2mm at the resting.
* New York Heart Association Class IV.
* Less than 45 days after myocardial infarction.
* Less than 3 months after acute heart failure.
* Patient has uncontrolled hypertension.
* Patient is pregnant.
* Patient has a medical condition that would limit study participation.
* Patient is enrolled in a concurrent study that may affect the outcome of this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianrong Zhao, MD, Principal Investigator — Ruijin Hospital Luwan Branch, Shanghai JiaoTong University School of Medicine; Jinbo Li, MD, Principal Investigator — Sixth People's Hospital Affiliated to Shanghai Jiaotong University
Locations (2):
- China (2):
  - Ruijin Hospital Luwan Branch, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality
  - Sixth People's Hospital Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen H, Zhao J, Zhou X, Li J, Wan Q, Huang J, Li H, Wu L, Yang S, Wang P. Impaired chronotropic response to physical activities in heart failure patients. BMC Cardiovasc Disord. 2017 May 25;17(1):136. doi: 10.1186/s12872-017-0571-9. PMID 28545575

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Case Group | Control Group
Started | 40 | 8
Completed | 40 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Case Group | Control Group | Total
Number analyzed (Participants) | 40 | 8 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (11.7) | 59.5 (3.2) | 55.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 30 | 5 | 35

OUTCOME MEASURES:

1. Primary Outcome: Chronotropic Incompetence Index of Patients With Heart Failure Disease
Description: Compare chronotropic incompetence index in patients with heart failure using an interventional diagnostic algorithm compared to standard of care diagnostics.
  Chronotropic Index = [achieved maximal HR-resting HR]/[age-predicted maximal HR-resting HR]. Normal CI is ~ 1 with low CI considered < 0.8
  Measurement described as: Chronotropic index=HRR/metabolic reserve.
Time Frame: Implant through 6 months
Population: Compare the case group for chronotropic incompetence using the interventional algorithm versus those in the control group.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Case Group | Control Group
Number analyzed (Participants) | 40 | 8
Index | 0.61 (0.11) | 0.72 (0.01)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline through 12 months follow-up.
Description: All cardiovascular AE's were collected.
Arm/Group | Case Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/8
Other Adverse Events (participants affected / at risk) | 0/40 | 0/8

LIMITATIONS AND CAVEATS:
Because the study was discontinued, none of objectives of the study were met, the pre-specified analyses for all objectives were not performed (per study protocol).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes